CLINICAL TRIAL: NCT02555618
Title: A Randomized Double-Blind Parallel-Group Comparative Phase 2 Study to Evaluate the Immunogenicity and Safety of a Single Subcutaneous Injection of TAK-850 in Comparison With Influenza HA Vaccine in Healthy Adult Subjects
Brief Title: Phase 2 Study of TAK-850 in Comparison With Influenza Hemagglutinin (HA) Vaccine in Healthy Adult Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TAK-850/CPH-003; U1111-1174-1290 (Registry Identifier: WHO); JapicCTI-153019 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-09-17; First posted 2015-09-21 (Estimated); Results first posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-11

CONDITIONS: Influenza Infection
Keywords: Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAK-850 (Experimental): A single dose of 0.5 mL TAK-850 (15 μg of hemagglutinin [HA] antigen per strain) is injected subcutaneously into the upper arm.
  Interventions: Biological: TAK-850
- Influenza HA Vaccine (Active Comparator): A single dose of the 0.5 mL influenza HA vaccine (15 μg of HA antigen per strain) is injected subcutaneously into the upper arm.
  Interventions: Biological: Influenza HA vaccine

INTERVENTIONS:
Biological: TAK-850 — TAK-850 subcutaneous injection
  Arms: TAK-850
Biological: Influenza HA vaccine — Influenza HA vaccine subcutaneous injection
  Arms: Influenza HA Vaccine

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of TAK-850 administered subcutaneously as a single dose versus influenza HA vaccination in an exploratory manner.

DETAILED DESCRIPTION:
This study is a phase 2, single dose study of TAK-850 (cell-culture derived TIV) administered subcutaneously in healthy Japanese adults, designed as a randomized, double-blind, parallel-group, comparative study to evaluate the immunogenicity and safety compared to an egg-derived TIV.

The drug being tested in this study is called TAK-850. TAK-850 was tested in healthy volunteers. This study looked at immunogenicity and safety of TAK-850 (cell-derived) compared to an egg-derived influenza vaccine.

The study enrolled 400 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the two groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* TAK-850
* Influenza HA vaccine All participants received one injection. This single center trial was conducted in Japan. The overall time to participate in this study was 22 days. Participants made multiple visits to the clinic, including a final visit 21 days after the vaccination for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator or subinvestigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written, informed consent form prior to the initiation of any study procedures.
3. The participant is a healthy Japanese adult male or female.
4. The participant is aged 20 to 49 years, inclusive, at the time of informed consent.
5. The participant has a body mass index (BMI) between 18.5 and 25.0 kg/m^2, inclusive, at the time of the eligibility evaluation.
6. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agreed to routinely use adequate contraception from signing of the informed consent throughout the duration of the study.

Exclusion Criteria:

1. The participant has received any investigational compound within 4 months prior to injection of study vaccine.
2. The participant has been vaccinated with seasonal influenza vaccine within 6 months prior to injection of study vaccine.
3. The participant has a history of influenza infection within 6 months prior to injection of study vaccine.
4. The participant has been vaccinated with TAK-850 before.
5. The participant is a study site employee, an immediate family member of such an employee, or in a dependent relationship with a study site employee who is involved in the conduct of this study (e.g., spouse, parent, child, sibling), or may consent under duress.
6. The participant has uncontrolled, clinically significant manifestations of neurological, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, endocrine, or other disorders, which may impact the ability of the participant to participate or potentially confound the study results.
7. The participant has an oral temperature >= 37.5 °C prior to injection of study vaccine on Day 1.
8. The participant has any medically diagnosed or suspected immune deficient condition.
9. The participant has an immune compromising condition or disease, or is currently undergoing a form of treatment or was undergoing a form of treatment that can be expected to influence immune response within 30 days prior to injection of study vaccine. Such treatments include systemic or high dose inhaled corticosteroids (> 800 µg/day of beclomethasone dipropionate or equivalent; the use of inhaled and nasal steroids that do not exceed this level will be permitted), radiation therapy, and other immunosuppressive and cytotoxic drugs.
10. The participant has received antipyretics within 4 hours prior to the injection of study vaccine.
11. The participant has a history of Guillain-Barré Syndrome, demyelinating disorders (including acute disseminated encephalomyelitis [ADEM] and multiple sclerosis), or convulsions.
12. The participant has a functional or surgical asplenia.
13. The participant has a rash, other dermatologic conditions, or tattoos which may interfere with the evaluation of injection site reaction.
14. The participant has a history of, or is infected with the Hepatitis B Virus (HBsAgs), Hepatitis C Virus (HCV), or Human Immunodeficiency Virus (HIV).
15. The participant has known hypersensitivity to any component of TAK-850 or Influenza HA Vaccine.
16. The participant has a history of severe allergic reactions or anaphylaxis.
17. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to injection of study vaccine or is unwilling to agree to abstain from excessive alcohol and drugs throughout the study.
18. The participant has received any blood products (blood transfusion or immunoglobulin) within 90 days prior to injection of study vaccine.
19. The participant has received a live vaccine within 4 weeks (28 days) or an inactivated vaccine within 2 weeks (14 days) prior to injection of study vaccine.
20. If female, the participant is pregnant or lactating or intending to become pregnant before signing of informed consent, during treatment, or within 12 weeks after injection of study vaccine; or intending to donate ova during this time period.
21. The participant has donated whole blood >= 200 mL within 4 weeks (28 days), >= 400 mL within 12 weeks (84 days), >= 800 mL within 52 weeks (364 days) or blood components within 2 weeks (14 days) prior to injection of study vaccine.
22. The participant has abnormal laboratory values that suggest a clinically significant underlying disease at the assessment prior to the injection of study vaccine, or the participant has the following laboratory abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) more than 3 times the respective upper limits of normal.
23. In the opinion of the investigator or subinvestigator, the participant is unlikely to comply with protocol requirements or is considered ineligible for any other reasons.

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 24 September 2015 to 18 November 2015.
Pre-assignment Details: Healthy Volunteers were enrolled equally in 1 of 2 groups, TAK-850 subcutaneous (SC) or Influenza hemagglutinin (HA) vaccine SC.
Period: Overall Study
Arm/Group | TAK-850 | Influenza HA Vaccine
Started | 200 | 200
Completed | 199 | 200
Not Completed | 1 | 0
Not completed — Sponsor's Circumstances | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAK-850 | Influenza HA Vaccine | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (9.61) | 31.5 (9.46) | 31.4 (9.52)
Age, Customized [Number; unit: participants]
  20 to 29 years | 102 | 98 | 200
  30 to 39 years | 46 | 47 | 93
  40 to 49 years | 52 | 55 | 107
Gender [Count of Participants; unit: Participants]
  Female | 94 | 95 | 189
  Male | 106 | 105 | 211
Region of Enrollment [Number; unit: participants]
  Japan | 200 | 200 | 400
Height [Mean (Standard Deviation); unit: cm] | 166.3 (8.41) | 166.0 (8.32) | 166.2 (8.35)
Weight [Mean (Standard Deviation); unit: kg] | 58.67 (8.918) | 57.69 (7.937) | 58.18 (8.445)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 21.10 (1.912) | 20.86 (1.752) | 20.98 (1.835)
Influenza Infection within 1 Year [Number; unit: participants]
  Yes | 14 | 11 | 25
  No | 186 | 189 | 375
Hemagglutination Inhibition (HI) Antibody Titer (Egg-derived)-A/H1N1 Strain [Number; unit: participants] — HI Antibody Titer data is only available for N=199, 200 respectively.
  participants
    Titer <40 | 74 | 65 | 139
    Titer ≥40 | 125 | 135 | 260
HI Antibody Titer (Egg-derived)-A/H3N2 Strain [Number; unit: participants] — HI Antibody Titer data is only available for N=199, 200 respectively.
  participants
    Titer <40 | 106 | 105 | 211
    Titer ≥40 | 93 | 95 | 188
HI Antibody Titer (Egg-derived)-B Strain [Number; unit: participants] — HI Antibody Titer data is only available for N=199, 200 respectively.
  participants
    Titer <40 | 93 | 98 | 191
    Titer ≥40 | 106 | 102 | 208

OUTCOME MEASURES:

1. Primary Outcome: Seroconversion Rate of Hemagglutination Inhibition (HI) Antibody Titer (Egg-Derived Antigen)
Description: Seroconversion rate was measured by hemagglutination inhibition (HI) antibody titer (egg-derived antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination.
  Seroconversion rate was defined as the percentage of participants achieving a minimal 4-fold increase from the Baseline HI antibody titer in participants with a Baseline titer ≥10, or achieving an HI antibody titer of ≥40 in participants with a Baseline titer <10.
Time Frame: Baseline and Day 22
Population: Full Analysis Set (FAS) included all randomized participants who received vaccination with study vaccine. 1 participant in the TAK-850 group discontinued the study before completion of the specified final observation and is excluded.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 | Influenza HA Vaccine
Number analyzed (Participants) | 199 | 200
percentage of participants
  A/H1N1 Strain | 47.7 [40.627 to 54.918] | 46.0 [38.948 to 53.172]
  A/H3N2 Strain | 31.2 [24.795 to 38.088] | 36.0 [29.350 to 43.071]
  B Strain | 28.6 [22.472 to 35.463] | 26.0 [20.068 to 32.658]
Statistical Analysis 1: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is difference of seroconversion rate between treatment groups for A/H1N1 Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to -20%; Rate difference = 1.7, 95% CI 2-sided [-7.983 to 11.415] — TAK-850 - Influenza HA Vaccine
Statistical Analysis 2: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is difference of seroconversion rate between treatment groups for A/H3N2 Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to -20%; Rate difference = -4.8, 95% CI 2-sided [-13.974 to 4.403] — TAK-850 - Influenza HA Vaccine
Statistical Analysis 3: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is difference of seroconversion rate between treatment groups for B Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to -20%; Rate difference = 2.6, 95% CI 2-sided [-6.082 to 11.320] — TAK-850 - Influenza HA Vaccine

2. Primary Outcome: Geometric Mean Titer (GMT) of HI Antibody Titer (Egg-Derived Antigen)
Description: Geometric mean titer (GMT) of HI antibody titer (egg-derived antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination. Day 1 data is reported for reference.
Time Frame: Days 1 and 22
Population: FAS included all randomized participants who received vaccination with study vaccine. 1 participant in the TAK-850 group discontinued the study before completion of the specified final observation and is excluded.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TAK-850 | Influenza HA Vaccine
Number analyzed (Participants) | 199 | 200
titer
  A/H1N1 Strain-Day 1 | 39.04 (5.256) [30.955 to 49.228] | 43.77 (4.794) [35.178 to 54.463]
  A/H1N1 Strain-Day 22 | 239.24 (3.098) [204.264 to 280.206] | 241.88 (2.839) [209.128 to 279.763]
  A/H3N2 Strain-Day 1 | 21.39 (4.558) [17.300 to 26.439] | 22.62 (4.823) [18.163 to 28.168]
  A/H3N2 Strain-Day 22 | 64.80 (4.643) [52.282 to 80.314] | 84.93 (5.496) [66.967 to 107.707]
  B Strain-Day 1 | 24.65 (3.898) [20.380 to 29.812] | 25.34 (4.211) [20.734 to 30.960]
  B Strain-Day 22 | 70.14 (3.652) [58.523 to 84.063] | 65.89 (4.197) [53.945 to 80.475]
Statistical Analysis 1: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is Geometric Mean Ratio between treatment groups for A/H1N1 Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to 0.5; Ratio of GMTs = 0.99, 95% CI 2-sided [0.7984 to 1.2253] — TAK-850/Influenza HA Vaccine
Statistical Analysis 2: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is Geometric Mean Ratio between treatment groups for A/H3N2 Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to 0.5; Ratio of GMTs = 0.76, 95% CI 2-sided [0.5544 to 1.0500] — TAK-850/Influenza HA Vaccine
Statistical Analysis 3: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is Geometric Mean Ratio between treatment groups for B Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to 0.5; Ratio of GMTs = 1.06, 95% CI 2-sided [0.8134 to 1.3931] — TAK-850/Influenza HA Vaccine

3. Secondary Outcome: Seroprotection Rate of HI Antibody Titer (Egg-Derived Antigen)
Description: Seroprotection rate, defined as the percentage of participants with HI antibody titer of ≥40, was measured by HI antibody titer (egg-derived antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination. Day 1 data is reported for reference.
Time Frame: Days 1 and 22
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 | Influenza HA Vaccine
Number analyzed (Participants) | 199 | 200
percentage of participants
  A/H1N1 Strain-Day 1 | 62.8 [55.697 to 69.543] | 67.5 [60.535 to 73.937]
  A/H1N1 Strain-Day 22 | 95.5 [91.589 to 97.911] | 97.0 [93.585 to 98.891]
  A/H3N2 Strain-Day 1 | 46.7 [39.645 to 53.921] | 47.5 [40.412 to 54.663]
  A/H3N2 Strain-Day 22 | 77.9 [71.477 to 83.451] | 78.0 [71.614 to 83.536]
  B Strain-Day 1 | 53.3 [46.079 to 60.355] | 51.0 [43.852 to 58.118]
  B Strain-Day 22 | 81.4 [75.295 to 86.558] | 76.0 [69.469 to 81.743]

4. Secondary Outcome: Geometric Mean Fold Increase in HI Antibody Titer (Egg-Derived Antigen)
Description: Geometric mean fold increase in HI antibody titer (egg-derived antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination, as compared with Baseline.
Time Frame: Baseline and Day 22
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | TAK-850 | Influenza HA Vaccine
Number analyzed (Participants) | 199 | 200
fold increase
  A/H1N1 Strain | 6.13 (5.496) [4.830 to 7.777] | 5.53 (5.353) [4.373 to 6.982]
  A/H3N2 Strain | 3.03 (4.268) [2.474 to 3.711] | 3.75 (4.861) [3.012 to 4.681]
  B Strain | 2.85 (3.399) [2.398 to 3.376] | 2.60 (3.356) [2.196 to 3.079]

5. Secondary Outcome: Seroconversion Rate of Single Radial Hemolysis (SRH) Antibody Titer (Egg-Derived Antigen)
Description: Seroconversion rate, defined as the percentage of participants with a Baseline SRH antibody titer of >4 mm^2 achieving a minimal 50% increase, or a Baseline SRH antibody titer of ≤4 mm^2 achieving a SRH antibody titer of ≥25 mm^2, as measured by single radial hemolysis (SRH) antibody titer (egg-derived antigen) for each of the three strains, 21 days after vaccination.
Time Frame: Baseline and Day 22
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 | Influenza HA Vaccine
Number analyzed (Participants) | 199 | 200
percentage of participants
  A/H1N1 Strain | 50.8 [43.591 to 57.894] | 44.0 [37.006 to 51.175]
  A/H3N2 Strain | 38.7 [31.890 to 45.839] | 47.5 [40.412 to 54.663]
  B Strain | 31.7 [25.262 to 38.611] | 34.0 [27.467 to 41.016]
Statistical Analysis 1: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is difference of seroconversion rate between treatment groups for A/H1N1 Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to -20%; Rate difference = 6.8, 95% CI 2-sided [-3.020 to 16.348]
Statistical Analysis 2: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is difference of seroconversion rate between treatment groups for A/H3N2 Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to -20%; Rate difference = -8.8, 95% CI 2-sided [-18.282 to 0.901]
Statistical Analysis 3: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is difference of seroconversion rate between treatment groups for B Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to -20%; Rate difference = -2.3, 95% CI 2-sided [-11.461 to 6.835]

6. Secondary Outcome: GMT of SRH Antibody Titer (Egg-Derived Antigen)
Description: GMT of SRH antibody titer (egg-derived antigen) for each of the three strains, 21 days after vaccination. Day 1 data is reported for reference.
Time Frame: Days 1 and 22
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mm^2
Arm/Group | TAK-850 | Influenza HA Vaccine
Number analyzed (Participants) | 199 | 200
mm^2
  A/H1N1 Strain-Day 1 | 32.4939 (2.98861) [27.88271 to 37.86773] | 33.7752 (2.85080) [29.18491 to 39.08753]
  A/H1N1 Strain-Day 22 | 83.6792 (1.70398) [77.67132 to 90.15189] | 79.9046 (1.46596) [75.75435 to 84.28212]
  A/H3N2 Strain-Day 1 | 23.6364 (2.99866) [20.27267 to 27.55832] | 24.8424 (2.79368) [21.52683 to 28.66874]
  A/H3N2 Strain-Day 22 | 48.0742 (2.03848) [43.51841 to 53.10687] | 53.5757 (1.87521) [49.07889 to 58.48463]
  B Strain-Day 1 | 45.6214 (2.00064) [41.40641 to 50.26551] | 46.3984 (1.89520) [42.44118 to 50.72466]
  B Strain-Day 22 | 74.3848 (1.32537) [71.51260 to 77.37238] | 75.8772 (1.32751) [72.93820 to 78.93464]
Statistical Analysis 1: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is Geometric Mean Ratio between treatment groups for A/H1N1 Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to 0.5; Ratio of GMTs = 1.05, 95% CI 2-sided [0.9559 to 1.1473] — TAK-850/Influenza HA Vaccine
Statistical Analysis 2: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is Geometric Mean Ratio between treatment groups for A/H3N2 Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to 0.5; Ratio of GMTs = 0.90, 95% CI 2-sided [0.7862 to 1.0241] — TAK-850/Influenza HA Vaccine
Statistical Analysis 3: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is Geometric Mean Ratio between treatment groups for B Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to 0.5; Ratio of GMTs = 0.98, 95% CI 2-sided [0.9273 to 1.0364] — TAK-850/Influenza HA Vaccine

7. Secondary Outcome: Seroprotection Rate of SRH Antibody Titer (Egg-Derived Antigen)
Description: Seroprotection rate, defined as the percentage of participants with SRH antibody titer ≥25 mm^2, was measured by SRH antibody titer (egg-derived antigen) for each of the three strains, 21 days after vaccination. Day 1 data is reported for reference.
Time Frame: Days 1 and 22
Population: FAS included all participants who received vaccination with study vaccine. 1 participant in the TAK-850 group discontinued the study before completion of the specified final observation and is excluded.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 | Influenza HA Vaccine
Number analyzed (Participants) | 199 | 200
percentage of participants
  A/H1N1 Strain-Day 1 | 70.4 [63.484 to 76.601] | 73.0 [66.285 to 79.020]
  A/H1N1 Strain-Day 22 | 97.0 [93.553 to 98.886] | 98.5 [95.679 to 99.690]
  A/H3N2 Strain-Day 1 | 63.8 [56.725 to 70.495] | 67.0 [60.017 to 73.470]
  A/H3N2 Strain-Day 22 | 89.4 [84.322 to 93.348] | 93.5 [89.141 to 96.494]
  B Strain-Day 1 | 87.9 [82.588 to 92.118] | 88.5 [83.245 to 92.569]
  B Strain-Day 22 | 99.5 [97.232 to 99.987] | 99.0 [96.435 to 99.879]

8. Secondary Outcome: Geometric Mean Fold Increase in SRH Antibody Titer (Egg-Derived Antigen)
Description: Geometric mean fold increase in SRH antibody titer (egg-derived antigen) for each of the three strains, 21 days after vaccination, as compared with Baseline.
Time Frame: Baseline and Day 22
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | TAK-850 | Influenza HA Vaccine
Number analyzed (Participants) | 199 | 200
fold increase
  A/H1N1 Strain | 2.5752 (2.83602) [2.22603 to 2.97921] | 2.3658 (2.88645) [2.04071 to 2.74262]
  A/H3N2 Strain | 2.0339 (2.54780) [1.78464 to 2.31798] | 2.1566 (2.44635) [1.90370 to 2.44314]
  B Strain | 1.6305 (1.81614) [1.49999 to 1.77232] | 1.6353 (1.77973) [1.50903 to 1.77222]

9. Secondary Outcome: Seroconversion Rate of HI Antibody Titer (Vero-Derived Antigen)
Description: Seroconversion rate, defined as the percentage of participants with a Baseline HI antibody titer of ≥10 achieving a minimal 4-fold increase, or a Baseline HI antibody titer of <10 achieving a HI antibody titer of ≥40, was measured by HI antibody titer (Vero-derived antigen) for each of the three strains, 21 days after vaccination.
Time Frame: Baseline and Day 22
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 | Influenza HA Vaccine
Number analyzed (Participants) | 199 | 200
percentage of participants
  A/H1N1 Strain | 40.2 [33.330 to 47.369] | 25.5 [19.614 to 32.128]
  A/H3N2 Strain | 27.1 [21.090 to 33.877] | 29.0 [22.816 to 35.819]
  B Strain | 19.6 [14.323 to 25.803] | 22.0 [16.464 to 28.386]
Statistical Analysis 1: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is difference of seroconversion rate between treatment groups for A/H1N1 Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to -20%; Rate difference = 14.7, 95% CI 2-sided [5.489 to 23.577]
Statistical Analysis 2: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is difference of seroconversion rate between treatment groups for A/H3N2 Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to -20%; Rate difference = -1.9, 95% CI 2-sided [-10.614 to 6.928]
Statistical Analysis 3: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is difference of seroconversion rate between treatment groups for B-Strain; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to -20%; Rate difference = -2.4, 95% CI 2-sided [-10.346 to 5.579]

10. Secondary Outcome: GMT of HI Antibody Titer (Vero-Derived Antigen)
Description: GMT of HI antibody titer (Vero-derived antigen) for each of the three strains, 21 days after vaccination. Day 1 data is reported for reference.
Time Frame: Days 1 and 22
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TAK-850 | Influenza HA Vaccine
Number analyzed (Participants) | 199 | 200
titer
  A/H1N1 Strain-Day 1 | 7.41 (2.395) [6.554 to 8.367] | 7.74 (2.346) [6.876 to 8.723]
  A/H1N1 Strain-Day 22 | 25.88 (4.297) [21.109 to 31.731] | 17.44 (3.978) [14.387 to 21.144]
  A/H3N2 Strain-Day 1 | 15.93 (3.549) [13.349 to 19.021] | 14.67 (3.722) [12.211 to 17.616]
  A/H3N2 Strain-Day 22 | 39.65 (4.449) [32.185 to 48.856] | 37.19 (5.313) [29.465 to 46.944]
  B Strain-Day 1 | 10.74 (2.826) [9.289 to 12.419] | 10.13 (2.721) [8.811 to 11.649]
  B Strain-Day 22 | 21.65 (4.004) [17.833 to 26.284] | 20.30 (3.770) [16.868 to 24.422]
Statistical Analysis 1: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is Geometric Mean Ratio between treatment groups for A/H1N1 Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to 0.5; Ratio of GMTs = 1.48, 95% CI 2-sided [1.1221 to 1.9623] — TAK-850/Influenza HA Vaccine
Statistical Analysis 2: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is Geometric Mean Ratio between treatment groups for A/H3N2 Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to 0.5; Ratio of GMTs = 1.07, 95% CI 2-sided [0.7806 to 1.4564] — TAK-850/Influenza HA Vaccine
Statistical Analysis 3: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is Geometric Mean Ratio between treatment groups for B Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to 0.5; Ratio of GMTs = 1.07, 95% CI 2-sided [0.8166 to 1.3934] — TAK-850/Influenza HA Vaccine

11. Secondary Outcome: Seroprotection Rate of HI Antibody Titer (Vero-Derived Antigen)
Description: Seroprotection rate, defined as the percentage of participants with HI antibody titer ≥40, was measured by HI antibody titer (Vero-derived antigen) for each of the three strains, 21 days after vaccination. Day 1 data is reported for reference.
Time Frame: Days 1 and 22
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 | Influenza HA Vaccine
Number analyzed (Participants) | 199 | 200
percentage of participants
  A/H1N1 Strain-Day 1 | 12.6 [8.298 to 17.984] | 11.0 [7.023 to 16.180]
  A/H1N1 Strain-Day 22 | 54.3 [47.079 to 61.334] | 40.0 [33.155 to 47.146]
  A/H3N2 Strain-Day 1 | 38.7 [31.890 to 45.839] | 32.0 [25.596 to 38.947]
  A/H3N2 Strain-Day 22 | 66.8 [59.827 to 73.331] | 60.0 [52.854 to 66.845]
  B Strain-Day 1 | 19.6 [14.323 to 25.803] | 22.0 [16.464 to 28.386]
  B Strain-Day22 | 43.2 [36.230 to 50.408] | 46.0 [38.948 to 53.172]

12. Secondary Outcome: Geometric Mean Fold Increase in HI Antibody Titer (Vero-Derived Antigen)
Description: Geometric mean fold increase in HI antibody titer (Vero-derived antigen) for each of the three strains, 21 days after vaccination, as compared with Baseline.
Time Frame: Baseline and Day 22
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | TAK-850 | Influenza HA Vaccine
Number analyzed (Participants) | 199 | 200
fold increase
  A/H1N1 Strain | 3.50 (4.066) [2.873 to 4.252] | 2.25 (3.539) [1.888 to 2.686]
  A/H3N2 Strain | 2.49 (3.584) [2.082 to 2.975] | 2.54 (3.593) [2.122 to 3.031]
  B Strain | 2.02 (3.046) [1.725 to 2.355] | 2.00 (2.831) [1.733 to 2.316]

13. Secondary Outcome: Seroconversion Rate of SRH Antibody Titer (Vero-Derived Antigen)
Description: Seroconversion rate, defined as the percentage of participants with a Baseline SRH antibody titer of >4 mm^2 achieving a minimal 50% increase, or a Baseline SRH antibody titer of ≤4 mm^2 achieving a SRH antibody titer of ≥25 mm^2, was measured by SRH antibody titer (Vero-derived antigen) for each of the three strains, 21 days after vaccination.
Time Frame: Baseline and Day 22
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 | Influenza HA Vaccine
Number analyzed (Participants) | 199 | 200
percentage of participants
  A/H1N1 Strain | 24.1 [18.352 to 30.677] | 23.0 [17.358 to 29.461]
  A/H3N2 Strain | 41.2 [34.294 to 48.385] | 42.0 [35.074 to 49.166]
  B Strain | 43.2 [36.230 to 50.408] | 40.0 [33.155 to 47.146]
Statistical Analysis 1: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is difference of seroconversion rate between treatment groups for A/H1N1 Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to -20%; Rate difference = 1.1, 95% CI 2-sided [-7.195 to 9.423] — TAK-850 - Influenza HA Vaccine
Statistical Analysis 2: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is difference of seroconversion rate between treatment groups for A/H3N2 Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to -20%; Rate difference = -0.8, 95% CI 2-sided [-10.369 to 8.803] — TAK-850 - Influenza HA Vaccine
Statistical Analysis 3: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is difference of seroconversion rate between treatment groups for B Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to -20%; Rate difference = 3.2, 95% CI 2-sided [-6.406 to 12.757] — TAK-850 - Influenza HA Vaccine

14. Secondary Outcome: GMT of SRH Antibody Titer (Vero-Derived Antigen)
Description: GMT of SRH antibody titer (Vero-derived antigen) for each of the three strains, 21 days after vaccination. Day 1 data is reported for reference.
Time Frame: Days 1 and 22
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TAK-850 | Influenza HA Vaccine
Number analyzed (Participants) | 199 | 200
titer
  A/H1N1 Strain-Day 1 | 7.4041 (2.32428) [6.58060 to 8.33056] | 7.7958 (2.26942) [6.95397 to 8.73955]
  A/H1N1 Strain-Day 22 | 16.2670 (2.13276) [14.63265 to 18.08382] | 15.2566 (2.32297) [13.56496 to 17.15930]
  A/H3N2 Strain-Day 1 | 19.7055 (2.07033) [17.79947 to 21.81561] | 19.1990 (2.14468) [17.26128 to 21.35415]
  A/H3N2 Strain-Day 22 | 32.4796 (1.76234) [30.00608 to 35.15703] | 33.2751 (1.85480) [30.52867 to 36.26852]
  B Strain-Day 1 | 28.2050 (2.17963) [25.29425 to 31.45059] | 28.2142 (2.23368) [25.22323 to 31.55982]
  B Strain-Day 22 | 52.1647 (1.53822) [49.11712 to 55.40139] | 49.7468 (1.55670) [46.76970 to 52.91348]
Statistical Analysis 1: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is Geometric Mean Ratio between treatment groups for A/H1N1 Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to 0.5; Ratio of GMTs = 1.07, 95% CI 2-sided [0.9106 to 1.2484] — TAK-850/Influenza HA Vaccine
Statistical Analysis 2: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is Geometric Mean Ratio between treatment groups for A/H3N2-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to 0.5; Ratio of GMTs = 0.98, 95% CI 2-sided [0.8686 to 1.0969] — TAK-850/Influenza HA Vaccine
Statistical Analysis 3: Comparison: TAK-850 vs Influenza HA Vaccine; The analysis is Geometric Mean Ratio between treatment groups for B Strain-Day 22; Test type: Non-Inferiority or Equivalence — Non inferiority margin is set to 0.5; Ratio of GMTs = 1.05, 95% CI 2-sided [0.9622 to 1.1427] — TAK-850/Influenza HA Vaccine

15. Secondary Outcome: Seroprotection Rate of SRH Antibody Titer (Vero-Derived Antigen)
Description: Seroprotection rate, defined as the percentage of participants with SRH antibody titer ≥25 mm^2, was measured by SRH antibody titer (Vero-derived antigen) for each of the three strains, 21 days after vaccination. Day 1 data is reported for reference.
Time Frame: Days 1 and 22
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 | Influenza HA Vaccine
Number analyzed (Participants) | 199 | 200
percentage of participants
  A/H1N1 Strain-Day 1 | 17.1 [12.132 to 23.048] | 13.0 [8.671 to 18.465]
  A/H1N1 Strain-Day 22 | 33.7 [27.140 to 40.692] | 33.0 [26.530 to 39.983]
  A/H3N2 Strain-Day 1 | 38.2 [31.411 to 45.328] | 42.5 [35.556 to 49.670]
  A/H3N2 Strain-Day 22 | 71.9 [65.065 to 77.990] | 74.0 [67.342 to 79.932]
  B Strain-Day 1 | 65.3 [58.272 to 71.917] | 65.5 [58.469 to 72.063]
  B Strain-Day 22 | 92.5 [87.872 to 95.720] | 93.5 [89.141 to 96.494]

16. Secondary Outcome: Geometric Mean Fold Increase in SRH Antibody Titer (Vero-Derived Antigen)
Description: Geometric mean fold increase in SRH antibody titer (Vero-derived antigen) for each of the three strains, 21 days after vaccination, as compared with Baseline.
Time Frame: Baseline and Day 22
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | TAK-850 | Influenza HA Vaccine
Number analyzed (Participants) | 199 | 200
fold increase
  A/H1N1 Strain | 2.1970 (2.03685) [1.98906 to 2.42676] | 1.9570 (2.16354) [1.75737 to 2.17938]
  A/H3N2 Strain | 1.6483 (1.71298) [1.52879 to 1.77705] | 1.7332 (1.71960) [1.60699 to 1.86926]
  B Strain | 1.8495 (1.91583) [1.6881 to 2.02546] | 1.7632 (2.03032) [1.59739 to 1.94618]

17. Secondary Outcome: Percentage of Participants With Solicited Local and Systemic Adverse Events (AEs)
Description: Participants recorded solicited injection site and systemic adverse events in a Subject Diary. Solicited Locals AEs were: Injection Site Pain, Injection Site Redness, Injection Site Swelling, Injection Site Induration and Injection Site Ecchymosis. Solicited Systemic AEs were: Pyrexia, Malaise, Chills, Fatigue, Headache, Sweaty, Myalgia, Arthralgia, Nausea and Vomiting.
Time Frame: 22 Days
Population: Safety Analysis Set included all participants who received vaccination with study vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-850 | Influenza HA Vaccine
Number analyzed (Participants) | 200 | 200
percentage of participants
  Injection site pain | 34.0 | 39.5
  Injection site redness | 23.5 | 28.0
  Injection site swelling | 15.5 | 20.0
  Injection site induration | 7.0 | 10.0
  Injection site ecchymosis | 3.5 | 4.5
  Pyrexia | 0.0 | 0.5
  Malaise | 10.5 | 11.0
  Chills | 2.5 | 4.5
  Fatigue | 10.5 | 6.5
  Headache | 7.0 | 9.0
  Sweaty | 0.5 | 1.5
  Myalgia | 3.5 | 5.5
  Arthralgia | 0.0 | 1.5
  Nausea | 1.5 | 2.0
  Vomiting | 0.5 | 1.0

18. Secondary Outcome: Percentage of Participants Reporting One or More Treatment-emergent Adverse Events (TEAE)
Description: Adverse events are defined as unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product, regardless of relationship to the medicinal product. TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: 22 days
Population: Safety Analysis Set included all participants who received vaccination with study vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-850 | Influenza HA Vaccine
Number analyzed (Participants) | 200 | 200
percentage of participants | 62.0 | 64.0

19. Secondary Outcome: Percentage of Participants With Abnormal Safety Laboratory Tests at Least Once Post Dose Reported as AEs
Description: The percentage of participants with any abnormal standard safety laboratory values (Chemistry, Hematology and Urinalysis) collected throughout the study reported as AEs.
Time Frame: 22 Days
Population: Safety Analysis Set included all participants who received vaccination with study vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-850 | Influenza HA Vaccine
Number analyzed (Participants) | 200 | 200
percentage of participants
  Blood creatine phosphokinase increased | 2.0 | 1.0
  Protein urine present | 0.5 | 0.5
  Blood bilirubin increased | 0.5 | 0.0
  Liver function test abnormal | 0.5 | 0.0
  White blood cell count increased | 0.5 | 0.0
  Alanine aminotransferase increased | 0.0 | 0.5
  Blood glucose increased | 0.0 | 0.5

ADVERSE EVENTS:
Time Frame: 22 Days
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-850 | Influenza HA Vaccine
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/200
Other Adverse Events (participants affected / at risk) | 117/200 | 122/200
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-850 (N=200) | Influenza HA Vaccine (N=200)
Injection site pain (General disorders) | 68 | 79
Injection site erythema (General disorders) | 47 | 56
Injection site swelling (General disorders) | 31 | 40
Injection site pruritus (General disorders) | 19 | 31
Injection site warmth (General disorders) | 17 | 29
Malaise (General disorders) | 21 | 22
Injection site induration (General disorders) | 14 | 20
Headache (Nervous system disorders) | 14 | 18
Fatigue (General disorders) | 21 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.